CLINICAL TRIAL: NCT02446054
Title: A Study to Evaluate the Effect of Musashino Diabetes Diet in Type II Diabetes Mellitus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celio Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013CMP-V2
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-05

CONDITIONS: Type II Diabetes Mellitus
Keywords: T2DM, type II diabetes Mellitus, HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One Arm Study (Experimental): provide Musashino T2DM diet for 12 weeks to T2DM patients, to evaluate the effect on glycosylated hemoglobin (HbA1c), progression and compliance during study period.
  Interventions: Dietary Supplement: Musashino T2DM diet

INTERVENTIONS:
Dietary Supplement: Musashino T2DM diet — provide Musashino T2DM diet for 12 weeks to T2DM patients, to evaluate the effect on glycosylated hemoglobin (HbA1c), progression and compliance during study period.

SUMMARY:
Evaluation the change of patients' glycosylated hemoglobin (HbA1c) after 12 weeks diet control

DETAILED DESCRIPTION:
In this study, we provide the delivery service of Musashino T2DM diet for 12 weeks to patients with T2DM, to evaluate the effect on glycosylated hemoglobin (HbA1c), progression and compliance during study period.

ELIGIBILITY:
Inclusion Criteria:

* A baseline of glycosylated hemoglobin(HbA1c) is, 10%≥HbA1c≥7%, during past 1 month
* The subject is able to understand and comply with protocol requirements, instrument
* The subject and/or subject's primary caregiver is able to have the telephone interview use computer and internet assess
* Signed and dated written informed consent

Exclusion Criteria:

* Pregnancy, breastfeeding or planning to become pregnant during the study
* Acute illness or infection requiring treatment within 14 days of study entry
* Other serious disease (e.g. Heart, lung, brain, liver) within 3 months
* Presence of malignancies
* Participate in other clinical trial within 30 days prior to this study
* Alcohol or drug abuse that would interfere with the ability to meet study requirements (opinion of investigator)
* Concurrent significant medical condition that would limit ability to participate in the study
* Consider by the investigator to be unsuitable for study participation, for any reason

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the change of glycosylated hemoglobin (HbA1c) | 12 weeks
  12 weeks diet control

SECONDARY OUTCOMES:
the change of patients' fasting blood Glucose | 12 weeks
the change of patients' fasting serum Insulin | 12 weeks
the change of patients' fasting serum C-peptide | 12 weeks
the change of EuroQol EQ-5D questionnaire | 12 weeks
the change of WHO-QoL questionnaire | 12 weeks
the patients' compliance questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CY Wang, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan

REFERENCES:
- [Background] 1.Saydah SH, Eberhardt MS, Loria CM, Brancati FL. Age and the burden of death attributable to diabetes in the United States. Am J Epidemiol 2002;156:714-9. 2. Pastors JG, Franz MJ, Warshaw H, Daly A, Arnold MS. How effective is medical nutrition therapy in diabetes care? J Am Diet Assoc 2003;103:827-31. 3. American Diabetes Association, Bantle JP, Wylie-Rosett J, Albright AL, et al. Nutrition recommendations and interventions for diabetes: a position statement of the American Diabetes Association. Diabetes Care 2008;31(Suppl 1):S61-78. 4. Robert E. Post, MD, MS, Arch G. Mainous III, PhD, Dana E. King, MD, MS, and Kit N. Simpson, DrPH Dietary Fiber for the Treatment of Type 2 Diabetes Mellitus: A Meta-Analysis J Am Board Fam Med 2012;25:16 -23.)